CLINICAL TRIAL: NCT01925521
Title: A phase1,Randomized,Double-blind,Placebo-controlled,Two-part,Sequential Ascending Single and Multiple Dose Study to Investigate the Safety, Tolerability and the PK and PD Profile of OPS-2071 in Healthy Male Korean Subjects
Brief Title: OPS-2071 Single and Multiple Dose Study to Investigate PK and PD Profile in Healthy Korean Male Subjects.
Acronym: OPS-2071Ph1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 341-KOA-1301i
Record Dates: First submitted 2013-08-12; First posted 2013-08-19 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Intestinal Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part1 : OPS-2071 (Experimental): Single dose, OPS-2071 30,60,120,240,300,600,900,1200mg/day
  Interventions: Drug: Part1 : OPS-2071
- Part1 : Placebo of OPS-2071 (Placebo Comparator): Single dose, Placebo
  Interventions: Drug: Part1 : Placebo of OPS-2071
- Part2 : OPS-2071 (Experimental): Multiple dose
  Interventions: Drug: Part2 : OPS-2071
- Part2 : Placebo of OPS-2071 (Placebo Comparator): Multiple doses, Placebo
  Interventions: Drug: Part2 : Placebo of OPS-2071

INTERVENTIONS:
Drug: Part1 : OPS-2071 — single oral dose under fasted condition
  Arms: Part1 : OPS-2071
Drug: Part1 : Placebo of OPS-2071 — single oral dose under fasted condition
  Arms: Part1 : Placebo of OPS-2071
Drug: Part2 : OPS-2071 — multiple twice-daily oral dosing for 5-7days
  Arms: Part2 : OPS-2071
Drug: Part2 : Placebo of OPS-2071 — multiple twice-daily oral dosing for 5-7days
  Arms: Part2 : Placebo of OPS-2071

SUMMARY:
The objective of this trial is to evaluate the safety and tolerability of single and multiple ascending oral doses of OPS-2071 in healthy male Korean

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a healthy male Korean aged 21 to 45 years, inclusive.
2. The subject has a body mass index (BMI) range of 18.5 to 25.0 kg/m2, inclusive, and weighs at least 50 kg.
3. The subject provided written, informed consent prior to any clinical study-specific procedures.
4. Male subject and his female spouse/partner who is of childbearing potential must be using highly effective barrier method of contraception starting at screening and continue throughout the clinical study period and for 3 months after final study drug administration.
5. Male subject must not donate sperm starting at screening and throughout the clinical study period and for 3 months after final study drug administration.

Exclusion Criteria:

1. Any clinically significant history of allergic conditions
2. Any history or evidence of any clinically significant disease or as judged by the Investigator.
3. Any clinically significant abnormality after the Investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or admission to the clinical unit.
4. A mean pulse of <45 or >90 beats per minute (bpm) and mean systolic blood pressure (SBP) >140 mmHg; mean diastolic blood pressure (DBP) >90 mmHg
5. A mean QTcB interval >450 ms at screening. If the mean QTcB exceeds the limits above, one additional triplicate ECG may be taken. If this triplicate also gives an abnormal result, the subject should be excluded.
6. Use of any prescribed or non-prescribed drugs in the 2 weeks prior to study drug administration, except for the occasional use of paracetamol (up to 2 g/day).
7. Consumption of grapefruit, pomelo, citrus fruits, starfruit, pomegranate, papaya, mango, rambutan, kiwi fruit, dragon fruit or passion fruit and products containing these fruits in the 2 weeks prior to study drug administration.
8. Excessive use of caffeine-containing beverages exceeding 500 mg caffeine/day (5 cups of coffee) and the inability to refrain from the use of caffeine-containing beverages during confinement in the clinical unit.
9. Current smokers and history of smoking within 3 months prior to screening.
10. History of drinking more than 21 units of alcohol per week (1 unit=10 g pure alcohol=250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to the first admission to the clinical unit.
11. Any use of drugs-of-abuse within 3 months prior to the first admission to the clinical unit.
12. Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.
13. Positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) 1 and/or 2 antibodies.
14. Participation in any clinical study within 3 months prior to the expected date of enrolment into the clinical study, provided that the clinical study did not entail a biological compound with a longer t½ or participation in more than 3 clinical studies within 12 months.
15. The subject has any other condition, which in the opinion of the Investigator precludes the subject's participation in the clinical study.
16. Employee of the Sponsor or the site.
17. Vulnerable subjects, e.g. subjects kept in detention.
18. Veins unsuitable for repeat venipuncture.
19. Are unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g. uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Part1 : adverse event, body weight, physical examination, vital sign, electrocardiogram, clinical laboratory test | 4days
Part2 : adverse event, body weight, physical examination, vital sign, electrocardiogram, clinical laboratory test, Bond and Lader visual analogue scale (BL VAS) | 21days
  Bond and Lader VAS: Day -1 and last dosing day (within 1 hour of expected Cmax)

SECONDARY OUTCOMES:
Part1 : Plasma pharmacokinetic parameters of OPS-2071 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
  Cmax, tmax, AUC and so on.
Part2 : Plasma Pharmacokinetic parameters of OPS-2071 | Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-morning-dose , Days 2 to 6: pre morning and evening dose, last dosing day: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose.
  Cmax, tmax, AUCtau, C12 and so on.
Part1 : Urine Pharmacokinetic parameter of OPS-2071 | Day 1: pre-dose, 0-4, 4-8, 8-12, 12-24, 24-48 and 48-72 hours post-dose
Part2 : Urine pharmacokinetic parameter of OPS-2071 | Day 1 and last dosing day : pre-morning dose, 0-4 post-morning dose, 4-8 post-morning dose and 8-12 hours post-morning dose.
Part1 : Fecal pharmacokinetic parameters of OPS-2071 | All post-dose samples
  Feces sample is collected in the 120-mg group only: All post-dose samples will be collected until discharge. Actual sampling time point will be recorded.
Part2 : Microflora test | Pre-dose, last dosing day to the day of discharge,. Day 21

CONTACTS AND LOCATIONS:
Overall Officials: InJin Jang, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea